CLINICAL TRIAL: NCT02740166
Title: Banding Ligation Plus Propranolol Versus Banding Ligation to Prevent Rebleeding of Esophageal Varices
Brief Title: Preventing Recurrent Bleeding After Eradication of Esophageal Varices
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Responsible Party: Principal Investigator, Wen-Chi Chen, Division of Gastroenterology and Hepatology, Kaohsiung Veterans General Hospital.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VGHKS13-CT6-06
Record Dates: First submitted 2016-04-12; First posted 2016-04-15 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-04

CONDITIONS: Esophageal Varices
Keywords: Esophageal Varices; propranolol; banding ligation
MeSH Terms: conditions — Esophageal and Gastric Varices | interventions — Propranolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Banding ligation group (No Intervention): Patients randomized to banding ligation group discontinue propranolol after eradication of esophageal varices.
- Propranolol group (Experimental): Patients randomized to propranolol group continue propranolol after eradication of esophageal varices.
  Interventions: Drug: propranolol

INTERVENTIONS:
Drug: propranolol — Patients randomized to propranolol group continue propranolol after eradication of esophageal varices.
  Arms: Propranolol group

SUMMARY:
Esophageal variceal bleeding is a severe complication of portal hypertension. Banding ligation plus non-selective beta-blockers is the current recommendation for prevention of recurrent bleeding. However, the optimal duration of use of non-selective beta-blockers is not well defined. This study aims at comparing the rebleeding rate and adverse effects in patients using or without using propranolol after eradication of esophageal varices.

DETAILED DESCRIPTION:
Cirrhotic patients with acute or recent esophageal variceal bleeding undergo banding ligation at 1-month interval until eradication of esophageal varices. Patients start propranolol (start with 30 mg daily) at 6th day after control of acute bleeding till eradication of esophageal varices, aiming at decreasing pulse rate to 25% or to 55 bpm while systolic pressure is above 85 mmHg. Patients randomized to propranolol group continue propranolol after eradication of esophageal varices. Patients randomized to banding ligation group discontinue propranolol after eradication of esophageal varices. Patients are followed to evaluate the incidence of rebleeding, adverse effects and survival.

ELIGIBILITY:
Inclusion Criteria:

* Age of 20 to 80 years
* Cirrhotic patients with acute or recent esophageal variceal bleeding proven by an endoscopy
* Stable hemodynamic condition for at least 3 days after banding ligation

Exclusion Criteria:

* Hepatocellular carcinoma or other malignancy
* Stroke or active sepsis
* Chronic kidney disease under renal replacement therapy
* Contraindications to non-selective beta-blockers
* A history of non-selective beta-blockers use, sclerotherapy, banding ligation, transjugular intrahepatic porto-systemic shunt, or shunt surgery
* Serum total bilirubin >10 mg/dL
* Grade III/IV hepatic encephalopathy
* Refractory ascites
* Hepato-renal syndrome
* Pregnancy
* Severe heart failure (NYHA Fc III/IV)
* Bronchial asthma or chronic obstructive pulmonary disease
* Second or third degree atrioventricular block
* Sick sinus syndrome
* Pacemaker use
* Severe hypotension
* Refusal to participate

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Estimated)
Dates: Start 2013-06; Primary Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
recurrent esophageal variceal bleeding | 6 years
  recurrent esophageal variceal bleeding after eradication of esophageal varices
mortality or liver transplantation | 6 years
  mortality or liver transplantation after eradication of esophageal varices

SECONDARY OUTCOMES:
adverse effects | 6 years
  adverse effects associated with non-selective beta-blockers and banding ligation

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Chi Chen, MD, Principal Investigator — Kaohsiung Veterans General Hospital.
Locations (1):
- Kaohsiung Veterans General Hospital, Kaohsiung City, Kaohsiung, Taiwan

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Gonzalez R, Zamora J, Gomez-Camarero J, Molinero LM, Banares R, Albillos A. Meta-analysis: Combination endoscopic and drug therapy to prevent variceal rebleeding in cirrhosis. Ann Intern Med. 2008 Jul 15;149(2):109-22. doi: 10.7326/0003-4819-149-2-200807150-00007. PMID 18626050
- [Background] Lo GH, Lai KH, Cheng JS, Chen MH, Huang HC, Hsu PI, Lin CK. Endoscopic variceal ligation plus nadolol and sucralfate compared with ligation alone for the prevention of variceal rebleeding: a prospective, randomized trial. Hepatology. 2000 Sep;32(3):461-5. doi: 10.1053/jhep.2000.16236. PMID 10960435
- [Background] de la Pena J, Brullet E, Sanchez-Hernandez E, Rivero M, Vergara M, Martin-Lorente JL, Garcia Suarez C. Variceal ligation plus nadolol compared with ligation for prophylaxis of variceal rebleeding: a multicenter trial. Hepatology. 2005 Mar;41(3):572-8. doi: 10.1002/hep.20584. PMID 15726659
- [Background] Kumar A, Jha SK, Sharma P, Dubey S, Tyagi P, Sharma BC, Sarin SK. Addition of propranolol and isosorbide mononitrate to endoscopic variceal ligation does not reduce variceal rebleeding incidence. Gastroenterology. 2009 Sep;137(3):892-901, 901.e1. doi: 10.1053/j.gastro.2009.05.049. Epub 2009 May 27. PMID 19481079
- [Derived] Chen WC, Yang TC, Lee PC, Wang YP, Hou MC, Lee FY. A Randomized Controlled Trial of Propranolol Use During Ligation Program for Secondary Prophylaxis of Esophageal Variceal Bleeding. Am J Gastroenterol. 2024 Feb 1;119(2):278-286. doi: 10.14309/ajg.0000000000002457. Epub 2023 Sep 11. PMID 37543755